CLINICAL TRIAL: NCT05841043
Title: A Multi-Center, Randomized, Double-masked, Vehicle-Controlled Phase III Clinical Study to Assess the Efficacy and Safety of SHR8028 Eye Drops for the Treatment of Dry Eye Disease
Brief Title: Efficacy and Safety of SHR8028 Eye Drops for the Treatment of Dry Eye Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SHR8028-301
Record Dates: First submitted 2023-04-24; First posted 2023-05-03 (Actual); Last update posted 2023-05-03 (Actual); Status verified 2023-04

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SHR8028 eye drops (Experimental)
  Interventions: Drug: SHR8028 eye drops
- Vehicle (Placebo Comparator)
  Interventions: Drug: Vehicle eye drops.

INTERVENTIONS:
Drug: SHR8028 eye drops — SHR8028 eye drops
  Arms: SHR8028 eye drops
Drug: Vehicle eye drops. — Vehicle eye drops.
  Arms: Vehicle

SUMMARY:
The study is being conducted to assess the efficacy, safety and tolerability of SHR8028 eye drops in comparison to the vehicle for the treatment of dry eye disease.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years old;
2. Provide written informed consent form;
3. Have a subject reported history of dry eye disease in both eyes for at least 180 days before the screening visit (visit 0);
4. Be currently (within 30 days before visit 0) using over-the-counter (OTC) eye drops, lubricating gels or tear neurostimulator device (such as True TearTM), and/or artificial tears for dry eye symptoms;
5. Have at least one eye meets criteria of moderate to severe dry eye both at visit 0&1
6. Be able and willing to follow instructions and participate in all study assessments and visits.

Exclusion Criteria:

1. Have any clinically significant slit-lamp findings at visit 0 that require treatment with prescription drugs and/or in the opinion of the investigator may interfere with study parameters, such as trauma, Stevens-Johnson syndrome, or advanced epithelial basement membrane disease;
2. Have dry eye disease secondary to scar formation, such as radiation, alkali burn, cicatricial pemphigus, and destruction of conjunctival goblet cells (i.e., destruction of conjunctival goblet cells caused by vitamin A deficiency);
3. Have active ocular allergy or ocular allergy that may occur during the study;
4. Be diagnosed with an ongoing ocular or systemic infection (bacterial, viral, or fungal), including fever, or be undergoing treatment with antibiotics at visit 0 and visit 1;
5. Be a woman who is pregnant, breastfeeding, or planning pregnancy;
6. Have an uncontrolled systemic disease;
7. Have allergies to investigational medicinal product (IMP) or its components: cyclosporin A or semi-fluorinated alkanes (SFA);
8. Be currently participating in other drug or device trials, or have used other investigational drugs or devices within 60 days before visit 0;
9. Have a condition which the investigator feels may put the subject at significant risk, may confound the study results, or may interfere with the subject's participation in the study significantly;
10. Have received or removed lacrimal duct embolism within 90 days before visit 0, or plan to receive or remove lacrimal duct embolism during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 206 (Actual)
Dates: Start 2021-03-04 (Actual); Primary Completion 2022-04-02 (Actual); Study Completion 2022-07-22 (Actual)

PRIMARY OUTCOMES:
Change in total corneal fluorescein staining (tCFS) score (National Eye Institute [NEI] scale) from baseline on Day 29 | Baseline, Day 29
Change in eye dryness score (visual analogue scale [VAS] Severity of Dryness) from baseline on Day 29 | Baseline, Day 29

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Peng R, Jie Y, Long Q, Gong L, Zhu L, Zhong X, Zhao S, Yan X, Gu H, Wu H, Li G, Zhang K, Krosser S, Xu R, Hong J. Water-Free Cyclosporine Ophthalmic Solution vs Vehicle for Dry Eye Disease: A Randomized Clinical Trial. JAMA Ophthalmol. 2024 Apr 1;142(4):337-343. doi: 10.1001/jamaophthalmol.2024.0101. PMID 38451509